CLINICAL TRIAL: NCT05462418
Title: Diathermy Versus Scalpel in the Transverse Abdominal Incision in Primigravida Obese Women Undergoing Cesarean Section
Brief Title: Diathermy vs Scalpel in Abdominal Incision in Women Undergoing CS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN2022-7
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Incision, Surgical
Keywords: Diathermy; scalpel; cesarean section; obese
MeSH Terms: conditions — Surgical Wound; Fever; Obesity | interventions — Electrosurgery; Diathermy; Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diathermy group (Active Comparator): Patients' incisions are completed using the unipolar diathermy from Whiteline until we reach the parietal peritoneum (cutting the Whiteline then coagulating until reaching the peritoneum). The used diathermy frequency was 50-70 MHz.
  Interventions: Procedure: electrosurgery
- scalpel (Active Comparator): patients had their incisions completed using the surgical scalpel till we reach the parietal peritoneum.
  Interventions: Procedure: scalpel

INTERVENTIONS:
Procedure: electrosurgery — incisions completed using use the unipolar diathermy from Whiteline till we reach the parietal peritoneum (cutting the Whiteline then coagulation till reaching the peritoneum). The used diathermy frequency was 50-70 MHz.
  Other Names: diathermy
  Arms: diathermy group
Procedure: scalpel — patients had their incisions completed using the surgical scalpel till we reach the parietal peritoneum.
  Arms: scalpel

SUMMARY:
Cesarean section is surging worldwide. For an extended period of surgical practice, the scalpel has been well-known as a gold-standard tool for making surgical incisions. The diathermy, electrocautery, is a substitute.

ELIGIBILITY:
Inclusion Criteria:

* Women with BMI 30- 40 Kg/m2.
* Women pregnant with singletons and planned to have a repeat elective lower-segment CS at 38-39 weeks' gestation due to having had one previous CS.
* Women pregnant with singletons and planned to deliver by lower-segment CS at 38-39 weeks' gestation for the first time (primi-section) due to obstetric indication.

Exclusion Criteria:

* Cases with coagulopathies eg. Hemophilia, von Willebrand disease
* Cases on anti-coagulant therapy eg. Heparin, warfarin
* Cases with chronic diseases expected to affect wound healing, such as diabetes, hypertension, liver diseases, chronic anemia, and renal impairment.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
blood loss | 30 min
  assess and compare intraoperative blood loss between both studied groups. This was done using visualization technique detecting numbers of fully soaked pads used during the incision.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Taymour, MD, Study Director — Cairo University
Locations (1):
- faculty of medicine - Cairo university, Cairo, Kasr El Ainy, Egypt

IPD SHARING:
Plan to Share IPD: No